CLINICAL TRIAL: NCT03988881
Title: Assessment of NOn-culprit Lesions With dobutamiNe Stress eChocardiography, compUted Tomography and Fractional fLow Reserve in Patients With Acute
Brief Title: DSE vs Invasive FFR vs CT-FFR
Acronym: NON-CULPRIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: Bajcsy-Zsilinszky Hospital (Other)
Responsible Party: Principal Investigator, Pál Maurovich-Horvat, associate professor, Semmelweis University Heart and Vascular Center
Other Study IDs: NON-CULPRIT
Record Dates: First submitted 2018-11-07; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Fractional Flow Reserve
Keywords: Dobutamine stress echocardiography; Fractional flow reserve; Computed tomography-fractional flow reserve; Non-culprit lesions; Myocardial infarction; Lesion specific ischemia
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 PCI Group: Patients after acute myocardial infarction and at least one moderate stenosis on the non-culprit vessels with positive dobutamine stress echocardiography and positive Fractional Flow Reserve recieving revascularization (PCI or CABG) Drug: Standard of care after acute myocardial infarction
  Interventions: Procedure: Revascularization
- Group 2 OMT group: Patients after acute myocardial infarction and at least one moderate stenosis on the non-culprit vessels with negative dobutamine stress echocardiography and negative Fractional Flow Reserve or the mismatching cases Standard of care after acute myocardial infarction

INTERVENTIONS:
Procedure: Revascularization — PCI or CABG
  Groups: 1 PCI Group

SUMMARY:
Data are limited regarding the optimal treatment of the non-culprit lesions (NCL) after myocardial infarction (MI). The NON-CULPRIT study is a prospective cohort study with a primary aim to compare invasive fractional flow reserve (FFR) and dobutamine stress echocardiography (DSE) for the evaluation and treatment of NCL in patients with MI.

As a secondary aim the investigators will assess the diagnostic performance of CT derived FFR as compared to invasive FFR and DSE measurements.

DETAILED DESCRIPTION:
Myocardial ischemia and coronary artery disease (CAD) burden both provide valuable prognostic information for adverse cardiac events. More than 50% of patients with acute myocardial infarction have multi-vessel coronary artery disease. However current evidence regarding the optimal treatment of the non-culprit lesions (NCL) after myocardial infarction (MI) is still limited.

The revascularization of NCL with at least moderate severity is associated with improved clinical outcomes, if significant ischemia was detected previously. Currently, there is no strict recommendation on the methods for detecting ischemia, therefore the current study aims to compare Dobutamine stress echocardiography (DSE) and invasive FFR for the evaluation and management of patients with MI and multi-vessel disease.

DSE and FFR measurements will be perfomed in patinets with at least one intermediate NCL. If both results are positive (new wall motion abnormality of at least two segments related to the examined coronary artery on DSE and FFR≤0,8 are declared as positive), stent implantation will be performed, if both results are negative or in case of mismatch, optimal medical treatment will be chosen.

Recent studies demonstrated the discrepancy between anatomical severity and hemodynamic relevance. Invasive fractional flow reserve (FFR) has emerged as the gold standard technique for the detection of lesion specific ischemia. The utilization of FFR in stable and acute chest pain patients can help in the selection of proper treatment strategy. The recently published Compare-Acute and DANAMI-Primulti trials have shown that in STEMI patients FFR-guided complete revascularization of NCL is beneficial as compared to infarct related lesion revascularization only.

However, in light of recent studies involving post-MI patients, invasive FFR might be limited for the assessment of NCL due to vessel remodeling, microvascular changes and altered hemodynamics.

Recent advancements in CT imaging allows for improved image quality and novel post-processing algorithms. Beyond anatomical data, functional information using coronary CT angiography (CTA) dataset and computational fluid dynamics simulations can be derived. CT derived FFR allows for the functional assessment of CAD in a non-invasive fashion.

Data regarding the diagnostic accuracy of CT-FFR as compared to other widely utilized functional tests are limited. Also, high-risk plaque features might affect lesion specific ischemia as detected by invasive FFR. Coronary CTA plus CT-FFR may help to identify patients requiring revascularization, even with controversial DSE and FFR results.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Moderate (40-80 %) stenosis of a non-culprit coronary artery
* Signed informed consent

Exclusion Criteria:

* Age under 18 years
* Age over 80 years
* Incurable malignant disease
* Patients for whom coronary CTA is contraindicated (History of severe and/or anaphylactic contrast reaction, severe renal insufficiency, inability to cooperate with scan acquisition and/or breathhold instructions)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who suffered acute MI and have at least one non/culprit leasion with a stenosis between 40-80%.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Acute myocardial infarction | From baseline to at least 2 years
  Detection of a rise and/or fall of cardiac biomarker values [preferably cardiac troponin (cTn)] with at least one value above the 99th percentile upper reference limit (URL) and with at least one of the following: Symptoms of ischaemia. New or presumed new significant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB).
Cardiovascular death | From baseline to at least 2 years
  Death occurs due to cardiovascular cause
Target vessel revascularization | From baseline to at least 2 years
  The Investigated Vessel needs Revascularisation due to angina

SECONDARY OUTCOMES:
Diagnostic performance of CT-FFR vs invasive FFR | From baseline to 3 months
  Diagnostic performance of CT-FFR as compared to invasive FFR
Diagnostic performance of CT-FFR vs DSE | From baseline to 3 months
  Diagnostic performance of CT-FFR as compared to DSE

CONTACTS AND LOCATIONS:
Overall Officials: Peter Andrassy, MD PhD, Principal Investigator — Bajcsy-Zsilinszky Hospital; Pal Maurovich-Horvat, MD PhD MPH, Study Director — Heart and Vascular Center, Semmelweis University
Locations (2):
- Hungary (2):
  - Bajcsy-Zsilinszky Hospital, Budapest, Pest County
  - Heart and Vascular Center, Semmelweis University, Budapest

IPD SHARING:
Plan to Share IPD: No
Data will be only shared with the pateints' other physicians

REFERENCES:
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Toth G, De Bruyne B, Casselman F, De Vroey F, Pyxaras S, Di Serafino L, Van Praet F, Van Mieghem C, Stockman B, Wijns W, Degrieck I, Barbato E. Fractional flow reserve-guided versus angiography-guided coronary artery bypass graft surgery. Circulation. 2013 Sep 24;128(13):1405-11. doi: 10.1161/CIRCULATIONAHA.113.002740. Epub 2013 Aug 28. PMID 23985788
- [Background] Toth G, Hamilos M, Pyxaras S, Mangiacapra F, Nelis O, De Vroey F, Di Serafino L, Muller O, Van Mieghem C, Wyffels E, Heyndrickx GR, Bartunek J, Vanderheyden M, Barbato E, Wijns W, De Bruyne B. Evolving concepts of angiogram: fractional flow reserve discordances in 4000 coronary stenoses. Eur Heart J. 2014 Oct 21;35(40):2831-8. doi: 10.1093/eurheartj/ehu094. Epub 2014 Mar 18. PMID 24644308
- [Background] De Rosa R, Piccolo R, Cassese S, Petretta A, D'Andrea C, D'Anna C, Piscione F, Chiariello M. Coronary flow reserve evaluation: basics, techniques and clinical applications. Minerva Cardioangiol. 2011 Dec;59(6):569-80. Epub 2009 Nov 30. PMID 19946255
- [Background] Corcoran D, Hennigan B, Berry C. Fractional flow reserve: a clinical perspective. Int J Cardiovasc Imaging. 2017 Jul;33(7):961-974. doi: 10.1007/s10554-017-1159-2. Epub 2017 Jun 2. PMID 28577046
- [Background] Rogers WJ, Bourassa MG, Andrews TC, Bertolet BD, Blumenthal RS, Chaitman BR, Forman SA, Geller NL, Goldberg AD, Habib GB, et al. Asymptomatic Cardiac Ischemia Pilot (ACIP) study: outcome at 1 year for patients with asymptomatic cardiac ischemia randomized to medical therapy or revascularization. The ACIP Investigators. J Am Coll Cardiol. 1995 Sep;26(3):594-605. doi: 10.1016/0735-1097(95)00228-v. PMID 7642848
- [Background] Hachamovitch R, Hayes SW, Friedman JD, Cohen I, Berman DS. Comparison of the short-term survival benefit associated with revascularization compared with medical therapy in patients with no prior coronary artery disease undergoing stress myocardial perfusion single photon emission computed tomography. Circulation. 2003 Jun 17;107(23):2900-7. doi: 10.1161/01.CIR.0000072790.23090.41. Epub 2003 May 27. PMID 12771008
- [Background] Shaw LJ, Berman DS, Maron DJ, Mancini GB, Hayes SW, Hartigan PM, Weintraub WS, O'Rourke RA, Dada M, Spertus JA, Chaitman BR, Friedman J, Slomka P, Heller GV, Germano G, Gosselin G, Berger P, Kostuk WJ, Schwartz RG, Knudtson M, Veledar E, Bates ER, McCallister B, Teo KK, Boden WE; COURAGE Investigators. Optimal medical therapy with or without percutaneous coronary intervention to reduce ischemic burden: results from the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial nuclear substudy. Circulation. 2008 Mar 11;117(10):1283-91. doi: 10.1161/CIRCULATIONAHA.107.743963. Epub 2008 Feb 11. PMID 18268144
- [Background] Brown OI, Clark AL, Chelliah R, Davison BJ, Mather AN, Cunnington MS, John J, Alahmar A, Oliver R, Aznaouridis K, Hoye A. Cardiogoniometry Compared to Fractional Flow Reserve at Identifying Physiologically Significant Coronary Stenosis: The CARDIOFLOW Study. Cardiovasc Eng Technol. 2018 Sep;9(3):439-446. doi: 10.1007/s13239-018-0354-1. Epub 2018 Apr 12. PMID 29651685
- [Background] Christou MA, Siontis GC, Katritsis DG, Ioannidis JP. Meta-analysis of fractional flow reserve versus quantitative coronary angiography and noninvasive imaging for evaluation of myocardial ischemia. Am J Cardiol. 2007 Feb 15;99(4):450-6. doi: 10.1016/j.amjcard.2006.09.092. Epub 2006 Dec 20. PMID 17293182
- [Background] Weidemann F, Jung P, Hoyer C, Broscheit J, Voelker W, Ertl G, Stork S, Angermann CE, Strotmann JM. Assessment of the contractile reserve in patients with intermediate coronary lesions: a strain rate imaging study validated by invasive myocardial fractional flow reserve. Eur Heart J. 2007 Jun;28(12):1425-32. doi: 10.1093/eurheartj/ehm082. Epub 2007 May 15. PMID 17504804
- [Background] Jung PH, Rieber J, Stork S, Hoyer C, Erhardt I, Nowotny A, Voelker W, Weidemann F, Ertl G, Klauss V, Angermann CE. Effect of contrast application on interpretability and diagnostic value of dobutamine stress echocardiography in patients with intermediate coronary lesions: comparison with myocardial fractional flow reserve. Eur Heart J. 2008 Oct;29(20):2536-43. doi: 10.1093/eurheartj/ehn204. Epub 2008 May 21. PMID 18499651